CLINICAL TRIAL: NCT07400250
Title: Phase II Study of Orelabrutinib in Combination With Romiplostim in Patients With Primary Immune Thrombocytopenia (ITP) Who Have Received at Least One Prior Line of Therapy
Brief Title: Phase II Study of Orelabrutinib in Combination With Romiplostim N01 in Patients With Primary Immune Thrombocytopenia (ITP) Who Have Received At Least One Prior Line of Therapy
Acronym: ORBIT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-ITP-II; InnoCare-ITP-001 (Other: InnoCare Pharma)
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: primary immune thrombocytopenia; orelabrutinib; romiplostim N01
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib combined with Romiplostim N01 (Experimental): The experimental arm will be treated orelabrutinib plus romiplostim N01. The study consists of three phases: 1) Core Treatment Phase (Weeks 1-24): Orelabrutinib 50mg orally once daily (fixed dose) + romiplostim N01 subcutaneously (starting dose 3ug/kg/week, administered once weekly). Platelet count and clinical symptoms are assessed weekly to adjust the dose of romiplostim N01 as appropriate, with a maximum dose of 10ug/kg/week. Patients with platelet count (PLT) <50×10⁹/L after 28 days of maximum-dose romiplostim N01 withdraw. 2) Tapering Phase (Weeks 25-32): Eligible patients (PLT ≥50×10⁹/L in the last two core phase visits) discontinue orelabrutinib, then taper romiplostim N01 (dose reduction + extended intervals); patients with two consecutive PLT <30×10⁹/L withdraw. 3) Follow-up Phase (Weeks 33-56): Successfully tapered patients are followed up every 4 weeks to monitor PLT and adverse events (graded per NCI-CTC AE 5.0).
  Interventions: Drug: Orelabrutinib; Drug: Romiplostim N01

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib will be given as 50mg per day orally, week 1-24
Drug: Romiplostim N01 — Core Treatment Phase Recommended starting dose: 3 μg/kg subcutaneously once weekly. Monitor platelet count (PLT) and symptoms weekly for dose adjustment, max 10 μg/kg/week. Therapeutic target: Maintain PLT within the range of 50-200×10⁹/L.
  1. PLT < 50×10⁹/L: Increase by 1-3 μg/kg/week to max dose. Discontinue study if PLT remains < 50×10⁹/L after 28d of max dose.
  2. 50-200×10⁹/L: Maintain the minimum effective dose to reduce bleeding risk.
  3. 200-400×10⁹/L: Decrease by 1-3 μg/kg/week. Discontinue if PLT ≥200×10⁹/L at 250 μg/week; resume when PLT <50×10⁹/L (extend interval if needed).
  4. PLT >400×10⁹/L: Suspend; resume at 1-3 μg/kg lower dose when PLT <200×10⁹/L (weekly monitoring).
  Tapering Phase For maintenance dose >3 μg/kg/week: Taper by 1-3 μg/kg/week to ≤3 μg/kg (250 μg/week), then extend intervals (weekly→every 10 days→every 2 weeks).
  1. PLT <30×10⁹/L: Maintain current dose.
  2. Two consecutive PLT <30×10⁹/L: Discontinue study.

SUMMARY:
To evaluate whether orelabrutinib combined with romiplostim N01 can improve the quality of remission, increase the probability of successful drug withdrawal, and prolong the time to treatment failure in patients with primary immune thrombocytopenia (ITP) who have received at least one line of prior therapy.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label Phase II study, enrolling adult patients with chronic primary immune thrombocytopenia (ITP) who failed first-line therapy. The study evaluates the efficacy and safety of orelabrutinib combined with romiplostim N01, focusing on the treatment regimen as follows:

* Core Treatment Phase (Weeks 1-24) Patients receive orelabrutinib 50mg orally once daily (fixed dose) and romiplostim N01 subcutaneously. Romiplostim N01 starts at 250ug/week (≈3ug/Kg) and is titrated within 1-10ug/Kg/week to maintain platelet count (PLT) at 50-200×10⁹/L. Dose adjustments: increase by 1-3ug/Kg/week if PLT <50×10⁹/L; decrease by 1-3ug/Kg/week if PLT 200-400×10⁹/L; suspend if PLT >400×10⁹/L. Patients with PLT <50×10⁹/L after 28 days of maximum-dose romiplostim N01 withdraw.
* Romiplostim N01 Tapering Phase (Weeks 25-32) Patients with PLT ≥50×10⁹/L in the last two core phase visits discontinue orelabrutinib. Romiplostim N01 is tapered: doses >3ug/Kg/week are reduced to 2-3ug/Kg/week, then dosing intervals extended (weekly→every 10 days→every 2 weeks). Patients with two consecutive PLT <30×10⁹/L withdraw.
* Follow-up Phase (Weeks 33-56) Successfully tapered patients are followed up every 4 weeks to monitor PLT and adverse events (graded per NCI-CTC AE 5.0). Relevant events are reported to the sponsor's Pharmacovigilance Department.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and provide written informed consent；
2. Age 18-80 years, inclusive, regardless of gender；
3. ECOG score 0 to 2；
4. Documented diagnosis of chronic primary Immune Thrombocytopenia (ITP) with a disease duration >12 months；
5. Patients with an inadequate sustained response, relapse, intolerance, or insufficient response to first-line ITP therapy (corticosteroids and/or intravenous immunoglobulin). Prior receipt of other ITP treatments is allowed, with no limit on the number of prior lines；
6. A history of response to prior standard ITP therapy (defined as achieving a platelet count ≥50×10⁹/L)；
7. During or following the most recent ITP treatment, patients must have experienced either: treatment failure (platelet count <30×10⁹/L after treatment, or failure to double the baseline count, or occurrence of bleeding), relapse after initial response (platelet count decreased to <30×10⁹/L, or fell below twice the baseline, or bleeding symptoms recurred), treatment intolerance, or an inability to maintain response after treatment discontinuation；
8. Subjects demonstrate adequate comprehension of and are able to comply with the study protocol requirements, and are willing to complete the study according to the schedule.

Exclusion Criteria:

1. Subjects suffer from severe ITP at screening;
2. Subjects have other diseases which mention in protocol;
3. Subjects develop intracranial hemorrhage within 6 months prior to screening;
4. Active and uncontrollable infection;

6. Subjects have a history of coagulopathy other than ITP; 7. Subjects with a history of malignancies; 8. History of major organ transplantation or hematopoietic stem cell/bone marrow transplantation; 9. Subjects with a known history of hypersensitivity to the investigational drug as described in the Protocol, or any ingredients; 10. Subjects with a Medication history and surgical history which mention in protocol; 11. Subjects do not meet the criterion of the laboratory test in protocol.

Withdrawal Criteria:

1. If, after 4 consecutive weeks of Romiplostim N01 administration at the maximum dose (10 µg/kg once weekly), the platelet count remains <50×10⁹/L and the investigator judges the investigational product to be ineffective for the subject, such that continued use is not in the subject's best interest；
2. Subjects who are unable to successfully undergo treatment tapering or discontinuation；
3. Subjects who, during the treatment period, require rescue therapy based on clinical assessment；
4. Subjects who withdraw their informed consent.
5. Occurrence of pregnancy during the trial period
6. Poor subject compliance or a significant protocol violation；
7. Loss to follow-up；
8. The investigator decides that withdrawal is necessary for the subject's safety；
9. Presence of other conditions, as determined by the investigator, that may affect the study results or lead to premature termination of the study；
10. Study completion or early termination of the entire study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
24-Week Sustained Platelet Response Rate | Up to 24 weeks
  The proportion of subjects with a platelet count (PLT) ≥ 50×10⁹/L in at least 4 out of the last 6 visits during the 24-week treatment period, without rescue therapy administered in the previous 4 weeks

SECONDARY OUTCOMES:
The sustained remission off-treatment (SROT) | Week 56
  At the end of follow-up (Week 56), the platelet count (PLT) is ≥ 30×10⁹/L and at least doubled compared to baseline, with no bleeding events and no rescue therapy administered during the period.
The cumulative number of weeks of platelet response | Up to 24 weeks
  Up to Week 24, the cumulative number of weeks with a platelet count (PLT) ≥ 50×10⁹/L
The time to first achievement of a platelet count ≥ 50×10⁹/L | Up to 24 weeks
  The time to first achievement of a platelet count ≥ 50×10⁹/L
Cumulative response time | Up to 24 weeks
  Number of cumulative weeks with platelet counts ≥ 30 × 10⁹/L and doubling of the baseline count and without bleeding by Week 24
Complete response rate | Up to 24 weeks
  The proportion of patients with a platelet count ≥ 100 × 10⁹/L on 3 consecutive visits at least 7 days apart and without bleeding
Time to First Rescue Therapy(TFRT) | Up to 24 Weeks
Bleeding Events | Up to 56 Weeks
  Assessed using the World Health Organization (WHO) Bleeding Scale. Clinically significant bleeding is defined and graded as follows:
  Grade 0 = No bleeding Grade 1 = Petechiae Grade 2 = Mild blood loss Grade 3 = Gross blood loss Grade 4 = Debilitating blood loss
Change From Baseline to Week 24 in ITP-PAQ Symptoms Score | Up to 24 Weeks
Treatment-emergent Adverse Events (TEAEs) | Up to 56 Weeks
  Common indicators include abnormalities in clinical symptoms and vital signs, as well as laboratory test abnormalities. The clinical manifestations, severity, time of onset, duration, management measures, and prognosis of these events are documented. The causal relationship to the investigational product(s) (Orelabrutinib or Ropylstimin N01) is assessed.
  Drug safety is evaluated according to the NCI-CTCAE version 5.0.
Exploratory Biomarkers | Up to 56 Weeks
  Including peripheral T/B cell subsets (including Th1, Th17, Th2, Treg, Breg).
Platelet membrane glycoprotein-specific antibodies; Cytokines: IL-4, IL-6, IL-17F, IL-9, IL-22, TGF-β, etc. | Up to 56 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tienan Zhu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China